CLINICAL TRIAL: NCT02412215
Title: Rotational Stability After Nanoflex Collamer Toric Intraocular Lens Implantation in Astigmatic Patients Undergoing Cataract Surgery
Brief Title: Rotational Stability After Nanoflex Collamer Toric Intraocular Lens Implantation in Astigmatic Patients
Acronym: T-IOL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Antonio Fea, Antonio Fea MD. PhD, University of Turin, Italy
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 0026769
Record Dates: First submitted 2015-03-29; First posted 2015-04-09 (Estimated); Last update posted 2015-04-09 (Estimated); Status verified 2015-04

CONDITIONS: Astigmatism
MeSH Terms: conditions — Astigmatism | interventions — Phacoemulsification

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Toric Nanoflex IOL (Experimental): Phacoemulsification with toric Nanoflex IOL implantation
  Interventions: Procedure: Phacoemulsification with toric Nanoflex IOL implantation; Device: NanoFlex toric Intraocular Lens

INTERVENTIONS:
Procedure: Phacoemulsification with toric Nanoflex IOL implantation — A self-sealing incision is made with a 2.2mm knife at 110°. Phacoemulsification is performed. The foldable nanoFlex toric IOL is injected in the capsular bag using the nanoPoint single-use injector system (STAAR) or 1620 sofTip Injector (ASICO). The IOL is rotated to align the cylinder axis with the steep corneal meridian using Z align function by Callisto Eye. Every movement of the IOL axis marks are noted.
Device: NanoFlex toric Intraocular Lens

SUMMARY:
This study aims to assess the rotational stability of the new collameric Nanoflex toric intraocular lens (T-IOL) by STAAR inserted in astigmatic patients after cataract surgery.

The purpose of this study is also to determine whether the use of a toric intraocular lens (T-IOL) improves visual acuity.

DETAILED DESCRIPTION:
A good rotational stability of toric intraocular lenses (T-IOL) allows an accurate refractive correction. However, many aspects -both pre-operative and post-operative- can interfere causing T-IOL rotation and misalignment.

Complete preoperative ocular evaluation is performed including slit-lamp examination, uncorrected distance visual acuity (UDVA), best-corrected visual acuity (BCVA), Javal keratometry, corneal Scheimplug tomography (Pentacam), optical biometry (IOL Master), Goldman applanation tonometry and fundus evaluation through dilated pupils. The spherical IOL power is calculated considering the axial length obtained with optical biometry, the magnitude of astigmatism derived from Javal keratometry and the steepest axis obtained with corneal tomography. The power of the toric IOL is determined with the online Staar Toric IOL calculator. The reference landmarks are also marked preoperatively with a sterile methylene blue fine point pen. The marking is rechecked in the operating theatre with the electronic toric marker ASICO.

Postoperative evaluation for IOL alignment and rotational stability is performed with slit-lamp photography on dilated pupils. Images are captured with Haag Streit slit lamp BQ 900 and are evaluated with the image-analysis software Protractor (Staar).

ELIGIBILITY:
Inclusion Criteria:

* Patients of 60 years of age ore more
* Cataract
* Corneal astigmatism of 1 diopter (D) or more

Exclusion Criteria:

* Primary or secondary pathological conditions of the cornea
* Zonular fibres pathologies (phacodonesis, pseudoexfoliation syndrome)
* Irregular astigmatism (corneal scar, keratoconus, pterygium)
* Traumatic cataract
* Previous ocular surgery
* Complications during cataract surgery

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-03; Primary Completion 2017-03 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Change in rotational stability of the toric intraocular lens (T-IOL). | Change of rotational stability at 1 day, 1 week, 1 month, 3 months, 6 months, 12 months and 18 months after surgery.
  The misalignment of the lens is defined as the difference (Δ) between the intended axis and the actual axis of the new collameric Nanoflex T-IOL by STAAR.

SECONDARY OUTCOMES:
Correction of the astigmatism. | Change in visual acuity at 1 day, 1 week, 1 month, 3 months, 6 months, 12 months and 18 months after surgery
  Effective correction evaluated through corrected distance visual acuity (CDVA) and uncorrected distance visual acuity (UDVA).

CONTACTS AND LOCATIONS:
Overall Officials: Antonio M Fea, MD, PhD, Principal Investigator — Department of Surgical Sciences, Ophthalmology Institute, University of Turin
Locations (1):
- Ophthalmology Institute, University of Turin, Turin, Italy

REFERENCES:
- [Background] Ferrer-Blasco T, Montes-Mico R, Peixoto-de-Matos SC, Gonzalez-Meijome JM, Cervino A. Prevalence of corneal astigmatism before cataract surgery. J Cataract Refract Surg. 2009 Jan;35(1):70-5. doi: 10.1016/j.jcrs.2008.09.027. PMID 19101427
- [Background] Rashad KM. Laser in situ keratomileusis for myopic astigmatism. J Refract Surg. 1999 Nov-Dec;15(6):653-60. doi: 10.3928/1081-597X-19991101-09. PMID 10590003
- [Background] Novis C. Astigmatism and toric intraocular lenses. Curr Opin Ophthalmol. 2000 Feb;11(1):47-50. doi: 10.1097/00055735-200002000-00007. PMID 10724827
- [Background] Chang DF. Early rotational stability of the longer Staar toric intraocular lens: fifty consecutive cases. J Cataract Refract Surg. 2003 May;29(5):935-40. doi: 10.1016/s0886-3350(02)01843-6. PMID 12781279
- [Background] Lane SS, Burgi P, Milios GS, Orchowski MW, Vaughan M, Schwarte E. Comparison of the biomechanical behavior of foldable intraocular lenses. J Cataract Refract Surg. 2004 Nov;30(11):2397-402. doi: 10.1016/j.jcrs.2004.03.041. PMID 15519095
- [Background] Lombardo M, Carbone G, Lombardo G, De Santo MP, Barberi R. Analysis of intraocular lens surface adhesiveness by atomic force microscopy. J Cataract Refract Surg. 2009 Jul;35(7):1266-72. doi: 10.1016/j.jcrs.2009.02.029. PMID 19545819
- [Background] Lane SS, Ernest P, Miller KM, Hileman KS, Harris B, Waycaster CR. Comparison of clinical and patient-reported outcomes with bilateral AcrySof toric or spherical control intraocular lenses. J Refract Surg. 2009 Oct;25(10):899-901. doi: 10.3928/1081597X-20090617-05. Epub 2009 Oct 12. PMID 19835331
- [Background] Koshy JJ, Nishi Y, Hirnschall N, Crnej A, Gangwani V, Maurino V, Findl O. Rotational stability of a single-piece toric acrylic intraocular lens. J Cataract Refract Surg. 2010 Oct;36(10):1665-70. doi: 10.1016/j.jcrs.2010.05.018. PMID 20870111
- [Background] Entabi M, Harman F, Lee N, Bloom PA. Injectable 1-piece hydrophilic acrylic toric intraocular lens for cataract surgery: efficacy and stability. J Cataract Refract Surg. 2011 Feb;37(2):235-40. doi: 10.1016/j.jcrs.2010.08.040. PMID 21241904
- [Background] Visser N, Bauer NJ, Nuijts RM. Toric intraocular lenses: historical overview, patient selection, IOL calculation, surgical techniques, clinical outcomes, and complications. J Cataract Refract Surg. 2013 Apr;39(4):624-37. doi: 10.1016/j.jcrs.2013.02.020. PMID 23522584
- [Background] Shimizu K, Misawa A, Suzuki Y. Toric intraocular lenses: correcting astigmatism while controlling axis shift. J Cataract Refract Surg. 1994 Sep;20(5):523-6. doi: 10.1016/s0886-3350(13)80232-5. PMID 7996408
- [Background] Till JS, Yoder PR Jr, Wilcox TK, Spielman JL. Toric intraocular lens implantation: 100 consecutive cases. J Cataract Refract Surg. 2002 Feb;28(2):295-301. doi: 10.1016/s0886-3350(01)01035-5. PMID 11821213
- [Background] Dick HB, Krummenauer F, Trober L. [Compensation of corneal astigmatism with toric intraocular lens: results of a multicentre study]. Klin Monbl Augenheilkd. 2006 Jul;223(7):593-608. doi: 10.1055/s-2006-926652. German. PMID 16855943
- [Background] Stewart CM, McAlister JC. Comparison of grafted and non-grafted patients with corneal astigmatism undergoing cataract extraction with a toric intraocular lens implant. Clin Exp Ophthalmol. 2010 Nov;38(8):747-57. doi: 10.1111/j.1442-9071.2010.02336.x. PMID 20497428
- [Background] Chang DF. Comparative rotational stability of single-piece open-loop acrylic and plate-haptic silicone toric intraocular lenses. J Cataract Refract Surg. 2008 Nov;34(11):1842-7. doi: 10.1016/j.jcrs.2008.07.012. PMID 19006728
- [Background] Alio JL, Agdeppa MC, Pongo VC, El Kady B. Microincision cataract surgery with toric intraocular lens implantation for correcting moderate and high astigmatism: pilot study. J Cataract Refract Surg. 2010 Jan;36(1):44-52. doi: 10.1016/j.jcrs.2009.07.043. PMID 20117704
- [Background] Bachernegg A, Ruckl T, Riha W, Grabner G, Dexl AK. Rotational stability and visual outcome after implantation of a new toric intraocular lens for the correction of corneal astigmatism during cataract surgery. J Cataract Refract Surg. 2013 Sep;39(9):1390-8. doi: 10.1016/j.jcrs.2013.03.033. Epub 2013 Jul 2. PMID 23827765
- [Background] Bascaran L, Mendicute J, Macias-Murelaga B, Arbelaitz N, Martinez-Soroa I. Efficacy and stability of AT TORBI 709 M toric IOL. J Refract Surg. 2013 Mar;29(3):194-9. doi: 10.3928/1081597X-20130129-02. PMID 23446016
- [Background] Chassain C. [Evaluation of visual performance after implantation of a double C-Loop toric intraocular lens]. J Fr Ophtalmol. 2014 Sep;37(7):507-13. doi: 10.1016/j.jfo.2014.02.007. Epub 2014 Aug 13. French. PMID 25127702
- [Background] Waltz KL, Featherstone K, Tsai L, Trentacost D. Clinical outcomes of TECNIS toric intraocular lens implantation after cataract removal in patients with corneal astigmatism. Ophthalmology. 2015 Jan;122(1):39-47. doi: 10.1016/j.ophtha.2014.06.027. Epub 2014 Nov 18. PMID 25444352
- [Background] Nguyen TM, Miller KM. Digital overlay technique for documenting toric intraocular lens axis orientation. J Cataract Refract Surg. 2000 Oct;26(10):1496-504. doi: 10.1016/s0886-3350(00)00442-9. PMID 11033397
- [Background] Rozema JJ, Gobin L, Verbruggen K, Tassignon MJ. Changes in rotation after implantation of a bag-in-the-lens intraocular lens. J Cataract Refract Surg. 2009 Aug;35(8):1385-8. doi: 10.1016/j.jcrs.2009.03.037. PMID 19631125
- [Background] Weinand F, Jung A, Stein A, Pfutzner A, Becker R, Pavlovic S. Rotational stability of a single-piece hydrophobic acrylic intraocular lens: new method for high-precision rotation control. J Cataract Refract Surg. 2007 May;33(5):800-3. doi: 10.1016/j.jcrs.2007.01.030. PMID 17466851
- [Background] Shah GD, Praveen MR, Vasavada AR, Rampal NV, Vasavada VA, Asnani PK, Pandita D. Software-based assessment of postoperative rotation of toric intraocular lens. J Cataract Refract Surg. 2009 Mar;35(3):413-8. doi: 10.1016/j.jcrs.2008.10.057. PMID 19251130
- [Background] Cha D, Kang SY, Kim SH, Song JS, Kim HM. New axis-marking method for a toric intraocular lens: mapping method. J Refract Surg. 2011 May;27(5):375-9. doi: 10.3928/1081597X-20101005-01. Epub 2010 Oct 15. PMID 20954592
- [Background] Sanders DR, Sarver EJ, Cooke DL. Accuracy and precision of a new system for measuring toric intraocular lens axis rotation. J Cataract Refract Surg. 2013 Aug;39(8):1190-5. doi: 10.1016/j.jcrs.2013.06.006. PMID 23889866
- [Background] Patel CK, Ormonde S, Rosen PH, Bron AJ. Postoperative intraocular lens rotation: a randomized comparison of plate and loop haptic implants. Ophthalmology. 1999 Nov;106(11):2190-5; discussion 2196. doi: 10.1016/S0161-6420(99)90504-3. PMID 10571358
- [Background] Chua WH, Yuen LH, Chua J, Teh G, Hill WE. Matched comparison of rotational stability of 1-piece acrylic and plate-haptic silicone toric intraocular lenses in Asian eyes. J Cataract Refract Surg. 2012 Apr;38(4):620-4. doi: 10.1016/j.jcrs.2011.10.037. Epub 2012 Jan 31. PMID 22296842
- [Background] Prinz A, Neumayer T, Buehl W, Vock L, Menapace R, Findl O, Georgopoulos M. Rotational stability and posterior capsule opacification of a plate-haptic and an open-loop-haptic intraocular lens. J Cataract Refract Surg. 2011 Feb;37(2):251-7. doi: 10.1016/j.jcrs.2010.08.049. PMID 21241906
- [Background] Mamalis N, Omar O, Veiga J, Tanner D, Pirayesh A, Fernquist DS. Comparison of two plate-haptic intraocular lenses in a rabbit model. J Cataract Refract Surg. 1996;22 Suppl 2:1291-5. doi: 10.1016/s0886-3350(96)80087-3. PMID 9051519
- [Background] Sacu S, Findl O, Linnola RJ. Optical coherence tomography assessment of capsule closure after cataract surgery. J Cataract Refract Surg. 2005 Feb;31(2):330-6. doi: 10.1016/j.jcrs.2004.04.057. PMID 15767154
- [Background] Kim MH, Chung TY, Chung ES. Long-term efficacy and rotational stability of AcrySof toric intraocular lens implantation in cataract surgery. Korean J Ophthalmol. 2010 Aug;24(4):207-12. doi: 10.3341/kjo.2010.24.4.207. Epub 2010 Aug 3. PMID 20714383
- [Background] Gomez-Bastar A, Jaimes M, Graue-Hernandez EO, Ramirez-Luquin T, Ramirez-Miranda A, Navas A. Long-term refractive outcomes of posterior chamber phakic (spheric and toric implantable collamer lens) intraocular lens implantation. Int Ophthalmol. 2014 Jun;34(3):583-90. doi: 10.1007/s10792-013-9860-1. Epub 2013 Oct 11. PMID 24114502